CLINICAL TRIAL: NCT06568887
Title: Effectiveness of 5% Dextrose Water (D/W) Versus Corticosteroid Injection for Pain Management of Sacroiliac Joint Dysfuntion
Brief Title: Effectiveness of 5% Dextrose Water Versus Corticosteroid Injection for Pain Management of SJD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MSRSW/Batch-Fall22/741
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Sacroiliac Joint Dysfunction
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextrose Water (Experimental)
  Interventions: Combination Product: Dextrose Water
- Corticosteroid Injection (Active Comparator)
  Interventions: Combination Product: Corticosteroid Injection

INTERVENTIONS:
Combination Product: Dextrose Water — Individuals in this group will receive three injections of 5% dextrose water per week for six weeks period to treat their pain in sacroiliac joint and then their responce will b documented.
  Arms: Dextrose Water
Combination Product: Corticosteroid Injection — Individuals in this group will receive three corticosteroid injections per week for a period of six weeks to treat their pain in Sacroiliac joint and then their responce will also be documented.
  Arms: Corticosteroid Injection

SUMMARY:
The sacroiliac joint (SIJ) is identified as a potential origin of low back pain and referred pain to the lower limb, with a prevalence rate ranging from 7% to 30%. Typically, SIJ pain manifests in the buttock and occasionally extends to the posterior aspect of the ipsilateral thigh, resembling pain originating from lumbar spine sources, such as the zygapophysial joints or intervertebral discs.

DETAILED DESCRIPTION:
For Sacroiliac Joint Dysfunction (SIJD) by examining the comparative effectiveness of two distinct interventions: the innovative 5% Dextrous Water (D/W) solution and the conventional corticosteroid injection. With corticosteroids associated with well-documented side effects and concerns about long-term use, the exploration of 5% D/W is particularly timely and holds promise as a potentially safer alternative.

ELIGIBILITY:
Inclusion Criteria:

* persons with SIJ pain for at least 3 months

Exclusion Criteria:

* Pregnancy or breastfeeding
* history of allergy or people contra indicated to our dose
* already received Corticosteroid injection in last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
VAS | 12 Months
  The Visual Analog Scale is a subjective measurement tool commonly used in research and clinical settings to assess the intensity or magnitude of various subjective characteristics or attitudes. It typically consists of a 100-mm horizontal or vertical line, with anchor points at each end representing extreme states (e.g., no pain to worst pain imaginable). Participants mark their perceived intensity on the line, and the distance from the starting point is measured to determine the score.
ODI | 12 months
  The Oswestry Disability Index is a widely used and well-established questionnaire designed to assess the impact of musculoskeletal conditions on an individual's daily activities and functionality, making it particularly relevant for conditions like piriformis syndrome. The questionnaire consists of ten sections addressing various aspects of daily life, including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling. Participants rate their level of disability in each section on a scale from 0 to 5, with 0 indicating no disability and 5 indicating maximum disability. The scores from each section are then summed and expressed as a percentage, with higher percentages representing greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No